CLINICAL TRIAL: NCT07126704
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Oral FB-101 in Healthy Adult Male Subjects
Brief Title: A Phase 1, SAD and MAD to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Oral FB-101 in Healthy Adult Male Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: 1ST Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FB101_P102
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- SAD 1. FB-101 10mg (Experimental)
  Interventions: Drug: FB-101; Drug: Placebo for FB-101
- SAD 2. FB-101 20mg (Experimental)
  Interventions: Drug: FB-101; Drug: Placebo for FB-101
- SAD 3. FB-101 40mg (Experimental)
  Interventions: Drug: FB-101; Drug: Placebo for FB-101
- MAD 4. FB-101 10mg QD (Experimental)
  Interventions: Drug: FB-101; Drug: Placebo for FB-101
- MAD 5. FB-101 20mg QD (Experimental)
  Interventions: Drug: FB-101; Drug: Placebo for FB-101
- MAD 6. FB-101 30mg QD (Experimental)
  Interventions: Drug: FB-101; Drug: Placebo for FB-101
- MAD 7. FB-101 10mg BID (Experimental)
  Interventions: Drug: FB-101; Drug: Placebo for FB-101
- MAD 8. FB-101 20mg BID (Experimental)
  Interventions: Drug: FB-101; Drug: Placebo for FB-101
- MAD 9. FB-101 30mg BID (Experimental)
  Interventions: Drug: FB-101; Drug: Placebo for FB-101

INTERVENTIONS:
Drug: FB-101 — FB-101 10mg
Drug: Placebo for FB-101 — Placebo for FB-101

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled study consisting of SAD and MAD investigation at a single clinical trial center conducted in healthy adult male subjects assessing the safety, tolerability, PK, and PD of oral FB-101 administration.

Up to 72 healthy adult male subjects will be enrolled. Additional subjects may be enrolled (8 subjects per cohort) if it is deemed appropriate following review (e.g., in the circumstances where a dose level is repeated, or an intermediate dose is conducted or to add another dose level(s) (higher than those planned)).

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy, adult, male 19-55 years of age, inclusive, at screening.
2. A continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to (the first) dosing and throughout the study, based on subject self-reporting.
3. Body mass index (BMI) ≥ 18.5 and ≤ 30.0 kg/m2 at screening.
4. Medically healthy with no clinically significant medical history, physical examination, neurological examination, ophthalmic examination, clinical laboratory profiles, vital signs, or safety 12-lead ECGs, as deemed by the PI or designee.
5. A non-vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days after (the last) dosing. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to (the first) dosing of the investigational product. A male who has been vasectomized less than 4 months prior to study (first) dosing must follow the same restrictions as a non-vasectomized male).
6. Must agree not to donate sperm from the first dosing until 90 days after the last dosing.
7. Able to swallow multiple capsules.

Key Exclusion Criteria:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. Is at suicidal risk in the opinion of the PI or designee.
4. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or pose an additional risk to the subject by their participation in the study.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number and severity of TEAEs | up to 2 month
  Number and severity of TEAEs following single ascending oral doses of FB-101 compared to placebo in healthy adult male subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea